CLINICAL TRIAL: NCT01049100
Title: Prospective, Randomised and Multi-centric Therapy Optimisation Study for Examining the Influence of Surgical Staging on the Oncological Results for Patients With Cervix Carcinoma of the FIGO Stages IIB-IV After Chemoradiation
Brief Title: Surgical Staging in Cervical Cancer Prior to Chemoradiation
Acronym: uterus11
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); Arbeitsgemeinschaft Radiologische Onkologie (Other)
Responsible Party: PD Dr. med. Simone Marnitz / Prof. Dr. med. Christhardt Köhler, Department of Radiooncology (Charité Campus Mitte und Virchow) / Department of Gynaecology (Charité Campus Mitte und Benjamin Franklin)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108771
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2009-08

CONDITIONS: Cervical Cancer
Keywords: Surgical Staging; Cervical Cancer; Chemoradiation; Outcome; Toxicity
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- operative staging (A) (Experimental): operative staging and systemic lymphadenectomy, paraaortal and pelvine, laparoscopic or open
  Interventions: Procedure: lymphadenectomy
- Standard (B) (No Intervention): No surgical intervention. Clinical Staging (FIGO) CT Abdomen / pelvic enlarged or suspicious lymphnodes--> CT controlled biopsy and histological analysis.
  Interventions: Other: Standard Staging

INTERVENTIONS:
Procedure: lymphadenectomy — paraaortal and pelvic lymphadenectomy laparoscopic or open
  Other Names: debulking, surgical staging
  Arms: operative staging (A)
Other: Standard Staging — clinical Staging (FIGO) (examination in narcosis, biopsy, cystoscopy, rectoscopy) X-Ray Radiograph of Thorax, Ultrasound of abdomen, CT abdomen / pelvis positive, suspicious lymphnodes--> CT controlled biopsy
  Other Names: FIGO Staging
  Arms: Standard (B)

SUMMARY:
The aim of this study is to determine whether the modified therapy on the basis of operative staging and systematic, pelvine and paraaortal lymphadenectomy for patients with cervical cancer of the FIGO stages IIB-IV prior to introducing radio-chemotherapy leads to a significant improvement of disease-free survival.

DETAILED DESCRIPTION:
The aim of this study is to determine whether the modified therapy on the basis of operative staging and systematic, pelvine and paraaortal lymphadenectomy for patients with cervical cancer of the FIGO stages IIB-IV prior to introducing radio-chemotherapy leads to a significant improvement of disease-free survival.

To this end, 250 patients with histologically verified cancer of the cervix uteri of the stages IIB-IV shall be randomised to a standard arm (ARM B), whereby the therapy shall be conducted on the basis of the clinical FIGO stage.

The patients randomised to the test arm (Arm A), after determining the clinical FIGO stage, shall initially receive an operative staging in the form of a pelvine paraaortal lymphadenectomy (laparoscopic or open). On the basis of the operatively obtained findings, a ("surgically") modified tumour stage shall be determined. This "surgical" tumour stage, which shall take into account the affection of the lymph nodes, the infiltration of the neighbouring organs and the intraperitoneal spread, shall serve as the basis for the execution of primary, combined radio-chemotherapy. The primary end-point is the disease-free survival of both groups, the secondary endpoints are overall survival, the local control of both groups, as well as the determination of toxicity and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky-Index =/> 70,
* age between 18 - 70 years
* histological assured cervical cancer (by biopsy)
* FIGO stages II B - IV
* written informed consent
* patient's ability to cooperate

Exclusion Criteria:

* neuroendocrine tumors or histological mixed types containing neuroendocrine fractions
* pregnancy, lactation,
* distant metastases, except paraaortal metastases
* other malignant diseases in anamnesis
* pelvic radiotherapy in anamnesis
* severe internal diseases
* psychiatric diseases which might query the trial attendance or follow-up
* HIV-Infection or AIDS
* drug addiction
* existing motoric or sensoric polyneuropathy > CTC Grad 1

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
DFS (disease-free survival) | 4 years

SECONDARY OUTCOMES:
OS, LC, QOL (overall survival, local control,quality of life, the determination of toxicity) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Simone Marnitz, PD, Study Chair — Department of Radiooncology (Charité Campus Mitte und Virchow), Charitéplatz 1, 10117 Berlin, Germany; Christhardt Köhler, Prof., Study Chair — Department of Gynaecology (Charité Campus Mitte und Benjamin Franklin), Charitéplatz 1, 10117 Berlin, Germany; Anja Dittgen, Principal Investigator — Department of Gynaecology (Charité Campus Mitte), Charitéplatz 1, 10117 Berlin, Germany
Locations (2):
- Germany (2):
  - Department of Gynaecology, Charité Campus Mitte und Benjamin Franklin, Berlin
  - Department of Radiooncology, Charité Campus Mitte und Campus Virchow, Berlin

REFERENCES:
- [Background] Sakuragi N. Up-to-date management of lymph node metastasis and the role of tailored lymphadenectomy in cervical cancer. Int J Clin Oncol. 2007 Jun;12(3):165-75. doi: 10.1007/s10147-007-0661-2. Epub 2007 Jun 27. PMID 17566838
- [Background] Subak LL, Hricak H, Powell CB, Azizi L, Stern JL. Cervical carcinoma: computed tomography and magnetic resonance imaging for preoperative staging. Obstet Gynecol. 1995 Jul;86(1):43-50. doi: 10.1016/0029-7844(95)00109-5. PMID 7784021
- [Background] Marnitz S, Kohler C, Roth C, Fuller J, Bischoff A, Wendt T, Schneider A, Budach V. Stage-adjusted chemoradiation in cervical cancer after transperitoneal laparoscopic staging. Strahlenther Onkol. 2007 Sep;183(9):473-8. doi: 10.1007/s00066-007-1675-4. PMID 17762920
- [Background] Bye A, Trope C, Loge JH, Hjermstad M, Kaasa S. Health-related quality of life and occurrence of intestinal side effects after pelvic radiotherapy--evaluation of long-term effects of diagnosis and treatment. Acta Oncol. 2000;39(2):173-80. doi: 10.1080/028418600430734. PMID 10859007
- [Background] Nag S, Erickson B, Thomadsen B, Orton C, Demanes JD, Petereit D. The American Brachytherapy Society recommendations for high-dose-rate brachytherapy for carcinoma of the cervix. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):201-11. doi: 10.1016/s0360-3016(00)00497-1. PMID 10924990
- [Background] Lai CH, Huang KG, Hong JH, Lee CL, Chou HH, Chang TC, Hsueh S, Huang HJ, Ng KK, Tsai CS. Randomized trial of surgical staging (extraperitoneal or laparoscopic) versus clinical staging in locally advanced cervical cancer. Gynecol Oncol. 2003 Apr;89(1):160-7. doi: 10.1016/s0090-8258(03)00064-7. PMID 12694671
- [Background] Denschlag D, Gabriel B, Mueller-Lantzsch C, Tempfer C, Henne K, Gitsch G, Hasenburg A. Evaluation of patients after extraperitoneal lymph node dissection for cervical cancer. Gynecol Oncol. 2005 Mar;96(3):658-64. doi: 10.1016/j.ygyno.2004.08.053. PMID 15721408
- See also: Association for Radiooncology — http://www.degro.org